CLINICAL TRIAL: NCT07170839
Title: Comparison of Eccentric and Combined Isotonic Exercises Combined With Extracorporeal Shock Wave Therapy in the Treatment of Lateral Epicondylitis
Brief Title: Combined Isotonic Exercise in the Treatment of Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, BÜŞRA CANDİRİ, assistant professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/103
Record Dates: First submitted 2025-08-19; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
Keywords: Pain, Exercise, Treatment, Extracorporeal shock wave therapy, Rehabilitation
MeSH Terms: conditions — Tennis Elbow; Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT Application (Experimental): A total of 5 sessions of ESWT were applied to all 3 groups, once a week for 5 weeks.
  Interventions: Other: ESWT Aplication
- Eccentric Treatment Protocol (Experimental): Patients in the eccentric exercise group underwent a protocol consisting of slow-progressive eccentric exercise of the wrist extensors combined with static stretching exercise, 3 times a week for 5 weeks.
  Interventions: Other: ECCENTRIC EXERCISE
- Combined Isotonic Exercise (Experimental): Patients in the combined isotonic exercise group underwent an eccentric-concentric exercise protocol combined with wrist isometric exercises 3 days a week for 5 weeks.
  Interventions: Other: COMBINED ISOTONIC EXERCISE

INTERVENTIONS:
Other: ESWT Aplication — All three groups received a total of five ESWT sessions, once a week for five weeks. All ESWT sessions were administered by the same physiotherapist, and the patients were positioned with their elbows flexed to 90 degrees and supported. ESWT was applied to sensitive points on the lateral epicondyle using a shock wave dose of 2000 pulses/session, with an intensity of 1.6 bar, a frequency of 10 Hz, and 1.6 bar. No analgesics or local anesthetics were administered before, during, or after the treatment.
  Arms: ESWT Application
Other: ECCENTRIC EXERCISE — Patients in the eccentric exercise group underwent a protocol consisting of slow-progressive eccentric wrist extensor exercises combined with static stretching exercises three times a week for 5 weeks. Eccentric exercises were performed without any resistance to eliminate gravity in the first week, and the intensity of the resistance was gradually increased using yellow elastic resistance bands in weeks 2-3 and red elastic resistance bands in weeks 4-5. Eccentric exercises were performed with the elbow extended, the forearm pronated, the wrist extended, and hanging down from the support surface. Patients were asked to slowly bend the wrist downward, count to 30, and then return to the starting position. Eccentric contractions were then performed in the same manner, and so on. Patients were instructed to continue the exercise if mild pain occurred but to stop the exercise if the pain increased to the point of preventing movement. Once patients tolerated the exercise, the lo
  Arms: Eccentric Treatment Protocol
Other: COMBINED ISOTONIC EXERCISE — Patients in the combined isotonic exercise group underwent an eccentric-concentric exercise protocol combined with wrist isometric exercises three days a week for 5 weeks. Similar to the eccentric training group, this group completed the training with resistance applied in the first week and elastic bands in subsequent weeks. In the first week, exercise training began with the patients' elbows in full extension, forearms in pronation, wrists in extension, and hanging from the support surface. Participants were asked to slowly bend their wrists for a count of 30, and the wrist extensors were eccentrically exercised. Immediately afterward, patients performed a concentric contraction while returning to the starting position (extension). Then, isometric contraction of the wrist extensors was maintained in the starting position for 30-45 seconds. Once the isometric contraction was achieved, concentric contraction continued, completing the exercise protocol.
  Arms: Combined Isotonic Exercise

SUMMARY:
This study was designed to investigate the effectiveness of the combined isotonic exercise technique applied with extracorporeal shock waves in the treatment of lateral epicondylitis.

Individuals aged 39-65 diagnosed with lateral epicondylitis were randomized using a sealed envelope method to one of the following groups: extracorporeal shock wave therapy, eccentric exercise and extracorporeal shock wave therapy, or combined isotonic exercise and extracorporeal shock wave therapy. Patients in the combined isotonic exercise and eccentric exercise groups were enrolled in a rehabilitation program under the supervision of a physiotherapist three days a week for five weeks. Extracorporeal shock wave therapy was also administered once a week for five weeks for all three groups. Pain intensity was assessed using the Visual Analog Scale, pressure pain threshold algometer, muscle strength using a hand-held dynamometer, grip strength using a digital hand-held dynamometer, and functionality using the Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lateral epicondylitis
* Having elbow pain lasting longer than 8 weeks
* Diagnosis of unilateral lateral epicondylitis
* Being a woman or man between the ages of 18 and 65
* No other lesions in or around the elbow

Exclusion Criteria:

* Cardiovascular, neurological, and neuromuscular diseases
* Prior trauma to the elbow area and previous elbow treatment
* Prior elbow surgery
* Peripheral nerve entrapment
* Corticosteroid injection within 6 months
* Bilateral elbow pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Baseline
  To determine patients' pain levels, pain intensity at rest and during activity was measured using a Visual Analog Scale (VAS). A 10-centimeter (cm) horizontal line was used on this scale, grading from "0: no pain" to "10: unbearable pain." Patients were asked to rate their current pain within this range.
Pain assessment | 5 weeks
  To determine patients' pain levels, pain intensity at rest and during activity was measured using a Visual Analog Scale (VAS). A 10-centimeter (cm) horizontal line was used on this scale, grading from "0: no pain" to "10: unbearable pain." Patients were asked to rate their current pain within this range.
Pressure Pain Assessment | Baseline
  An algometer was used to measure the pressure pain threshold. The 1-cm tip of the device was placed perpendicular to the patient's arm, with the arm in 30 degrees of abduction and the elbow in 90 degrees of flexion, and the forearm and wrist supported. The patient was asked to report the first time the applied pressure produced pain. This value was recorded on an assessment form in kg/cm².
Pressure Pain Assessment | 5 weeks
  An algometer was used to measure the pressure pain threshold. The 1-cm tip of the device was placed perpendicular to the patient's arm, with the arm in 30 degrees of abduction and the elbow in 90 degrees of flexion, and the forearm and wrist supported. The patient was asked to report the first time the applied pressure produced pain. This value was recorded on an assessment form in kg/cm².
Muscle Strength Assessment | Baseline
  Wrist extensor and middle finger muscle strength were measured using a hand-held dynamometer (Lafayette Instrument®, Lafayette, UK). The device was placed on the lateral surface of the metacarpal bones while the forearm was resting on the support surface. Participants were asked to perform an isometric contraction against the device in the direction of wrist extension for 5 seconds. The measured values were recorded on an evaluation form. Middle finger extension strength was tested with both the forearm and hand resting on the support surface.
Muscle Strength Assessment | 5 weeks
  Wrist extensor and middle finger muscle strength were measured using a hand-held dynamometer (Lafayette Instrument®, Lafayette, UK). The device was placed on the lateral surface of the metacarpal bones while the forearm was resting on the support surface. Participants were asked to perform an isometric contraction against the device in the direction of wrist extension for 5 seconds. The measured values were recorded on an evaluation form. Middle finger extension strength was tested with both the forearm and hand resting on the support surface.
Grip Strength Measurement | Baseline
  A Baseline digital handheld dynamometer (300 LB / 135 KG®) was used to measure maximum grip strength in patients. For this measurement, patients were asked to sit upright in a chair. With the arm and shoulder in a neutral position, the elbow in 90-degree flexion, the forearm in neutral, the wrist in slight extension, and ulnar deviation, the patient was instructed to squeeze the dynamometer firmly. The measured value was recorded in kilograms (kg). Three repetitions were performed for the affected hand, with a 1-minute rest period between repetitions. Grip strength was objectively measured by averaging these three values.
Grip Strength Measurement | 5 weeks
  A Baseline digital handheld dynamometer (300 LB / 135 KG®) was used to measure maximum grip strength in patients. For this measurement, patients were asked to sit upright in a chair. With the arm and shoulder in a neutral position, the elbow in 90-degree flexion, the forearm in neutral, the wrist in slight extension, and ulnar deviation, the patient was instructed to squeeze the dynamometer firmly. The measured value was recorded in kilograms (kg). Three repetitions were performed for the affected hand, with a 1-minute rest period between repetitions. Grip strength was objectively measured by averaging these three values.
Determining the Functionality Level | Baseline
  The Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH), developed for use in upper extremity musculoskeletal disorders, was used to determine patients' functional levels and symptoms. This questionnaire consists of three sections and 30 questions. Twenty-one questions address difficulties experienced by patients related to activities, five address disease symptoms, and the remaining questions assess work, sleep, social function, and patient self-confidence.
Determining the Functionality Level | 5 weeks
  The Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH), developed for use in upper extremity musculoskeletal disorders, was used to determine patients' functional levels and symptoms. This questionnaire consists of three sections and 30 questions. Twenty-one questions address difficulties experienced by patients related to activities, five address disease symptoms, and the remaining questions assess work, sleep, social function, and patient self-confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- İnönü Üniversitesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhabra G, Wang A, Ebert JR, Edwards P, Zheng M, Zheng MH. Lateral Elbow Tendinopathy: Development of a Pathophysiology-Based Treatment Algorithm. Orthop J Sports Med. 2016 Nov 1;4(11):2325967116670635. doi: 10.1177/2325967116670635. eCollection 2016 Nov. PMID 27833925
- [Background] Wilps T, Kaufmann RA, Yamakawa S, Fowler JR. Elbow Biomechanics: Bony and Dynamic Stabilizers. J Hand Surg Am. 2020 Jun;45(6):528-535. doi: 10.1016/j.jhsa.2020.01.016. Epub 2020 Apr 13. PMID 32299691
- [Result] Marshall NR, Randell MR, Nicholls AJ. Elbow anatomy, biomechanics and clinical examination. Shoulder Elbow. 2024;16(2):81-88.